CLINICAL TRIAL: NCT04918524
Title: The Clinical Features and Pregnancy Outcomes of Patients With Connective Tissue Disease :a Prospective Cohort Study
Brief Title: The Clinical Features and Pregnancy Outcomes of CTD Patients
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Chief Physician, Qilu Hospital of Shandong University
Other Study IDs: CTD with Pregnancy QiluH
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Connective Tissue Diseases; Pregnancy Related
Keywords: Connective tissue disease; Pregnancy outcomes; Clinical features; Risk factors
MeSH Terms: conditions — Connective Tissue Diseases | interventions — Prednisone; prednylidene; Hydroxychloroquine; Aspirin; Agouti Signaling Protein; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Antiphospholipid syndrome (APS): The cohort includes that patients who meet the proposed Sydney criteria.
  Interventions: Drug: Prednisone; Drug: Hydroxychloroquine; Drug: Aspirin; Drug: low molecular weight heparin Enoxaparin
- Undifferentiated connective tissue disease (UCTD): The cohort includes the patients who are diagnosed with UCTD: at least one presence of auto-antibodies, including antinuclear antibody (ANA), anti-extractable nuclear antigen (ENA) antibodies, anti-doublestranded DNA (ds-DNA) antibody, antiphospholipid antibodies (aPL), and non-criteria aPL (NC-aPL), with at least one symptoms or signs suggesting CTD ,while not fulfilling any classification criteria of a defined CTD.
  Interventions: Drug: Prednisone; Drug: Hydroxychloroquine; Drug: Aspirin; Drug: low molecular weight heparin Enoxaparin

INTERVENTIONS:
Drug: Prednisone — 5-30mg, po, once per day(Qd) prescribed if needed and adjusted due to patient response
  Other Names: Pred
Drug: Hydroxychloroquine — 100-200mg, po, twice per day (Bid) prescribed if needed and adjusted due to patient response.
  Other Names: HCQ
Drug: Aspirin — 100mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response to 32 weeks of pregnancy. 75mg po, once per day (Qd) to 34 weeks of pregnancy. 50mg po, once per day (Qd) to 36 weeks of pregnancy.
  Other Names: Asp
Drug: low molecular weight heparin Enoxaparin — 40-60mg, ih, Subcutaneous injection, once per day (Qd) or twice per day (Bid) if needed and adjusted due to patient response.
  Other Names: LMWH

SUMMARY:
Connective tissue disease (CTD) is a common group of autoimmune diseases, mainly including systemic lupus erythematosus (SLE), antiphospholipid syndrome (APS) , and so on. APS is caused by autoimmune disorders that cause recurrent miscarriage, thrombosis, and thrombocytopenia, and often secondary to connective tissue diseases such as SLE. Undifferentiated connective tissue disease (UCTD) is currently considered to be an independent disease in the classification of CTD. And women of childbearing age who suffer UCTD is more common than that in other definite CTDs. Therefore, the impact of the disease flare and the influence of medicine on pregnancy and lactation are important for these patients who may suffer high-risk of abnormal pregnance.

DETAILED DESCRIPTION:
Objective: To study the risk factors of poor pregnancy outcomes in CTD patients, and evaluate impact of different therapies on the maternal and fetal health.

Methods: Our department and Shanghai Gothic Network Technology Co.Ltd. jointly established the chronic disease management of CTD patients during pregnancy and lactation by using Smart System of Disease Management (SSDM). With this platform, patients in pregnancy can consult with rheumatologists face to face and follow-up regularly.

Follow-up: Consultation and followup will be scheduled every 4 weeks from confirmed pregnancy until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women who meet the following inclusion criteria will be eligible to participate in the study:

  1. Age between 20-45 years;
  2. Diagnosed with APS: patients meet the Sydney classification criteria;
  3. Diagnosed with UCTD: at least one presence of auto-antibodies, including antinuclear antibody (ANA), anti-extractable nuclear antigen (ENA) antibodies, anti-doublestranded DNA (ds-DNA) antibody, antiphospholipid antibody(aPL), and non-criteria aPL (NC-aPL), with at least one symptoms or signs suggesting connective tissue disease(CTD) , while not fulfilling any classification criteria of a defined CTD.
  4. Participate voluntarily in this study, willing to use medication and follow-up according to treatment plan, and sign informed consent.

Exclusion Criteria:

* Women who meet any of the following criteria will be excluded from the study:

  1.Any known etiology of previous pregnancy loss:
  1. Known paternal, maternal or embryo chromosome abnormality.
  2. Maternal endocrine dysfunction: corpus luteal insufficiency; polycystic ovarian syndrome; premature ovarian failure (follicle stimulating hormone, FSH ≥20uU/L in follicular phase);
  3. hyperprolactinemia; diabetes mellitus; other hypothalamic pituitary-adrenal axis abnormality
  4. Maternal anatomical abnormality: uterine malformation; Asherman syndrome; cervical incompetence; uterine fibrosis more than 5 cm.Vaginal infection.
  5. Any known severe cardiac, hepatic, renal, hematological or endocrinal diseases:

  2. Any active infection: Active infection including V aricella zostervirus(VZV), human immunodeficiency virus (HIV), Human papillomavirus (HPV),syphilis or tuberculosis.

  3. Allergic to prednisone, hydroxychloroquine, low-molecular-weight heparin or aspirin.

  4.Disease history as follows:
  1. Past history of digestive ulcers or upper gastrointestinal hemorrhage.
  2. Past history of malignancy.
  3. Past history of epilepsia or psychotic disorders.

  5.Women have been diagnosed with Systemic lupus erythematosus

  6. Women who disagree or cannot complete pregnancy and follow-up after delivery.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female with pregnance in accordance with the diagnostic criteria of connective tissue disease
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | After 28 weeks of gestation
  Percentage of all patients that lead to live birth after 28 weeks of gestation

SECONDARY OUTCOMES:
Early fetal loss | within 10 weeks of gestation
  Spontaneous pregnancy loss within 10 weeks of gestation
Late fetal loss | after 10 weeks of gestation
  Spontaneous pregnancy loss after 10 weeks of gestation
Stillbirth | after 20 weeks of gestation
  Spontaneous pregnancy loss after 20 weeks of gestation
Preterm delivery | between 28 and 37 weeks of gestation
  Live birth before 37 weeks of gestation
Low-weight birth | after 28 weeks of gestation
  newborns with low weight (<2500g)
Premature rupture of membranes | after 28 weeks of gestation
  the number of participants complicated with premature rupture of membranes
Placental abruption | after 28 weeks of gestation
  the number of participants complicated with placental abruption
Fetal growth retardation (FGR) | after 12 weeks of gestation
  weight below the 10th percentile for the gestational age
Number of participants with low amniotic fluid during pregnancy | after 12 weeks of gestation
  the number of participants whose B-ultrasound indicates low amniotic fluid during pregnancy
Number of participants with abnormal S / D values during pregnancy | after 12 weeks of gestation
  the number of participants whose B-ultrasound indicates abnormal S / D values during pregnancy
Number of participants with placental hematoma during pregnancy | during pregnancy, an average of 10 months
  the number of participants whose B-ultrasound indicates placental hematoma during pregnancy
Eclampsia | after 20 weeks of gestation
  New-onset hypertension after 20 weeks of gestation, with or without proteinuria > 300mg/24h, with or without any organ damage with seizures
Gestational diabetes | through study completion, an average of 10 months
  the number of participants who were diagnosed with gestational diabetes
Gestational hypertension | through study completion, an average of 10 months
  the number of participants who were diagnosed with gestational hypertension
Number of participants with placental infarction | at delivery
  the number of participants whose placenta with infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Yang, Dr., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No